CLINICAL TRIAL: NCT05172778
Title: Observational Study of the Performance of Cephen Reagents in the Context of Research Into Lupus Anticoagulants
Acronym: LA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8246
Record Dates: First submitted 2021-11-23; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Lupus Anticoagulant
Keywords: Lupus Anticoagulant; Coagulation; Phospholipid
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lupus anticoagulants (are antiphospholipid antibodies (PSA), the screening of which is done by demonstrating prolongation of coagulation times corrected by the intake of phospholipids (PL).

Learned societies (ISTH, CLSI) thus recommend, for the research of LA, to carry out initially two screening tests with a low concentration in PL: a time of diluted Russell viper venom (DRVVT) as well as a time activated partial thromboplastin (TCA). If one of these screening tests is positive, it is recommended to perform a second confirmation test using the same principle (DRVVT or TCA) and containing a higher concentration of PL.

The current LA screening method at the Hematology Laboratory of Strasbourg University Hospital includes: a pair of DRVVT screening / confirmation (STA-Staclot DRVV Screen and Confirm, Diagnostica Stago, France) and a screening TCA (PTT-A , Diagnostica Stago, France).

This study aims to compare with the current method of the investigators a pair of TCA screening / confirmation (Cephen LS / Cephen, Hyphen Biomed, France).

ELIGIBILITY:
Inclusion criteria:

* Major subject
* blood sample already analyzed in the laboratory as part of the treatment by the reference method
* Patient who did not express his opposition to the reuse of his data and his blood sample for the technical study.

Exclusion criteria:

* Minor patient
* Patient under curatorship, guardianship or legal protection
* Patient who expressed his opposition to the use of his data
* Insufficient sample

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject with blood sample already analyzed in the laboratory as part of the treatment by the reference method
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Observational study of the performance of Cephen reagents in the context of research into lupus anticoagulants | Files analysed retrospectively from January 01, 2019 to December 31, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Agathe HERB, PharmD, Principal Investigator — Laboratoire d'Hématologie - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Laboratoire d'Hématologie - Hôpitaux Universitaires de Strasbourg, Strasbourg, France